CLINICAL TRIAL: NCT05764967
Title: Comparative Effects Of Low Dye Taping Technique And Temporary Felt Insoles On Pain And Disability In Children With Pes Planus
Brief Title: Low Dye Taping Technique and Temporary Felt Insoles on Pain and Disability in Children With Pes Planus.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/22/0746
Record Dates: First submitted 2023-01-04; First posted 2023-03-13 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Pes Planus
Keywords: Disability; Insoles; Low Dye Taping; Pain; Pes Planus
MeSH Terms: conditions — Flatfoot; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Dye Taping (Experimental): One Arm will be given Low Dye taping. The augmented low-Dye technique, involves applying a device consisting of a spur and mini-stirrups to the foot and then adding reverse sixes and calcaneal slings to an anchor on the distal one-third of the leg. A rigid 38-mm sports tape with zinc oxide adhesive will be used for all of the taping procedures. Prior to application of the tape, any hair in the region will be shaved and the foot and leg will be washed with soap and warm water to remove any dirt or oils that might decrease the adhesion of the tape. The Transverse Tibial Rotation (TTR) measurements will be repeated following application of tape.
  Interventions: Other: Low Dye Taping
- Temporary Felt Insoles (Active Comparator): other will be given temporary shoe insoles. A temporary orthosis will be fabricated from 7-mm orthopedic felt. The orthosis consist of two parts, a medial longitudinal buttress and a navicular/sustentaculum tali pad. The medial longitudinal buttress will extend from the posterior calcaneus to the first metatarsal head and from the medial border of the foot to the bisection of the calcaneus and calcaneal recess will be cut out. A navicular/sustentaculum tali pad will extend from the sustentaculum tali to the cuneiform.
  Interventions: Other: Temporary Felt Insoles

INTERVENTIONS:
Other: Low Dye Taping — The augmented low-Dye technique, involves applying a device consisting of a spur and mini-stirrups to the foot and then adding reverse sixes and calcaneal slings to an anchor on the distal one-third of the leg. A rigid 38-mm sports tape with zinc oxide adhesive is used for all of the taping procedures.
  Arms: Low Dye Taping
Other: Temporary Felt Insoles — A temporary orthosis is fabricated from 7-mm orthopedic felt.The subject stands on his or her template while the TTR pointer is attached to the medial tibial plateau of the leg using a Velcro strap. An outline of the position of the device on the tibial plateau is drawn onto the skin with an indelible ink pen to allow for accurate relocation between all trials. TTR is measured in relaxed calcaneal stance while the subject wearing shoes. Measurements are recorded onto a data-collection sheet. Each measurement performes twice. The subject are given orthosis inserted into the shoe. All shoes are visually assessed to ensure that they will not induce pronation or internal rotation.
  Arms: Temporary Felt Insoles

SUMMARY:
This study aims to determine comparative effects of low dye taping technique and temporary felt insoles on pain and disability in children with pes planus.

DETAILED DESCRIPTION:
Pes planus is a foot arch deformity, is also known as flexible flat foot. Foot arch plays an important role in cushioning ground impact and stabilizing the body in standing and walking. Children with pes planus lack an elastic foot arch to attenuate the impact force. This condition results in pain and impaired lower limb function. Low Dye taping and shoe insoles are used to treat Pes Planus. Low Dye taping technique is designed to off-load the plantar fascia and provide medial ankle arch support. It is a classic taping method incorporating functional mechanical support of the foot and ankle. Low-Dye taping is commonly used to support the longitudinal and transverse arches of the foot.

A shoe insole is the footbed or material inside the shoe that the bottom or plantar surface of your foot lays on. In most well-made shoes today, the material or insole is removable. There are shoes that have glued in insoles, however in general these are shoes that are not as well made. The removable insoles that come in most shoes vary in type and material ranging from very simple thin cushioning to sophisticated multiple layered arch support inserts. The aim of this study is to compare the effects of Low dye taping and shoe insoles on pain and disability in children with pes planus.

The study will be Randomized Clinical trial. Total twenty four subjects will be assigned randomly by using block randomization into two groups (12 in each group). Both Groups will be experimental groups. Group A will be given low dye taping and Group B would be given temporary felt insoles. After confirmation of diagnosis with medical history and physical examination as well as different movement palpation tests and pain provocation tests are recommended. The Foot and Ankle Ability Measure (FAAM) and Numeric Pain Rating Scale (NPR) would be used as an outcome measure tools for pain and disability respectively. Measure will be taken at (Baseline and at the end of treatment session). The collected data will be analyzed in Statistical Package for the Social Sciences (SPSS) 27.0. Parametric/non-parametric tests will be applied after testing normality of data.

ELIGIBILITY:
Inclusion Criteria:

* 6-12year
* vertical navicular height of 10 mm or more
* A Vernier height gauge (Mitutoyo Corp, Tokyo, Japan) calibrated to 0.02 mm was used to measure vertical navicular height.

Exclusion Criteria:

* current injuries to the lower extremities that had required a reduction in activity levels and/or treatment by a health-care practitioner.
* severe orthopedic or neurologic conditions, and a known allergy to sports tape.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-04-05 (Actual)

PRIMARY OUTCOMES:
Foot And Ankle Ability Measure- FAAM | 2 months
  A self-report outcome tool that was created to evaluate physical function in people with foot and ankle-related disabilities. This Questionnare consists of 29 items which is subdivided into two sub-scales: the Foot and Ankle Ability Measure, Activities of Daily Living (ADL) Subscale having 21 items and the Foot and Ankle Ability Measure, Sports Subscale having 8 items.
Numeric Pain Rating Scale- NPRS | 2 months
  It is an outcome measure that provides a one-dimensional assessment of pain severity. It is an 11-point numeric scale spans from "0" to "10," with "pain as awful as you can conceive" or "worst pain imaginable" denoting one extreme of pain and "no pain" denoting the other.
Low Dye Taping Technique (To overcome pain and disability) | 2 months
  it is designed to off-load the plantar fascia and provide medial ankle arch support. It is a classic taping method incorporating functional mechanical support of the foot and ankle
Temporary Felt Insoles (To overcome pain and disability) | 2 months
  the inner sole of a shoe or boot. a loose additional inner sole used to give extra warmth, comfort.

CONTACTS AND LOCATIONS:
Overall Officials: Arnab Altaf, Mphill, Principal Investigator — Riphah International University
Locations (1):
- Children Hospital Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No